CLINICAL TRIAL: NCT04833985
Title: Intracardiac Versus Transesophageal Echocardiography Versus Fluoroscopy Only Guidance for Combined Catheter Ablation for Atrial Fibrillation and Left Atrial Appendage Occlusion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: xieruiqin (Other)
Responsible Party: Sponsor-Investigator, xieruiqin, director of cardiology department, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEE vs.ICE vs.fluoroscopy only
Record Dates: First submitted 2021-03-29; First posted 2021-04-06 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2020-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- transesophageal echocardiography guidance (Experimental)
  Interventions: Procedure: LAAC combined with radiofrequency ablation
- intracardiac echocardiography guidance (Experimental)
  Interventions: Procedure: LAAC combined with radiofrequency ablation
- fluoroscopy only guidance (Experimental)
  Interventions: Procedure: LAAC combined with radiofrequency ablation

INTERVENTIONS:
Procedure: LAAC combined with radiofrequency ablation — Each patient received the same group of patients with simple radiofrequency ablation and LAAC

SUMMARY:
A total of 75 patients with atrial fibrillation were scheduled to receive left atrial appendage occlusion combined with radiofrequency ablation, which were divided into 3 groups. The operation was performed under the guidance of intracardiac echocardiography and transesophageal echocardiography and fluoroscope only respectively (allocation ratio 1:1:1). During the operation, the total amount of contrast medium injected, the fluoroscopy time and the time from femoral vein puncture to transseptal puncture to closure were recorded in all patients. All patients underwent transesophageal echocardiography before and 3 months after operation, and the results were explained by two experienced ultrasound doctors to measure the presence of left atrial thrombus, residual shunt and device-related thrombus. All patients were examined by transthoracic echocardiography 3 months after operation to evaluate new pericardial effusion, pericardial tamponade, instrument embolization / displacement and so on. The baseline clinical and surgical features and hospitalization outcomes of patients guided by ICE and TEE and fluoroscopy only were recorded and compared. Clinical endpoints include death, new pericardial effusion that does not require pericardiocentesis, tamponade with pericardiocentesis, instrument embolism / displacement, bleeding at the entry site, thromboembolic events (stroke / transient ischemic attack [TIA]). The purpose of this study was to evaluate the feasibility, safety and effectiveness of intracardiac echocardiographic (ICE)-guided and transesophageal echocardiographic (TEE)-guided and fluoroscopy only-guided left atrial appendage occlusion combined with radiofrequency ablation. The average follow-up time is 3 months.

ELIGIBILITY:
Inclusion Criteria:

AF attack occurred in patients with a duration of more than one year, patients taking class I and class III antiarrhythmic drugs could not prevent AF, patients younger than 80 years old Cha2ds2-vasc score ≥2 and HAS-BLED score ≥3, not suitable for long-term oral anticoagulant drugs.

Exclusion Criteria:

Patients with a history of atrial thrombosis or valvular heart disease (moderate or severe valve stenosis or severe valve regurgitation), patients undergoing prosthetic heart valve replacement, pregnant women, patients with previous liver and kidney diseases, malignant tumors or blood system diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
injected contrast media | in the procedure
  milliliter
fluoroscopy time were recorded | in the procedure
  mGy

SECONDARY OUTCOMES:
the time from femoral vein puncture to transseptal puncture to closure were recorded | in the procedure
  second
The size of the LAA | in the procedure
  millimeter
the size of the selected umbrella in operation | in the procedure
  millimeter
residual shunt and DRT after transcatheter closure of left atrial appendage detected | before operation and 3 months after operation
  Transesophageal echocardiography
new pericardial effusion were detected | 3 months after operation
  Transthoracic echocardiography
pericardial tamponade were detected | 3 months after operation
  Transthoracic echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China